CLINICAL TRIAL: NCT04557241
Title: Brief Informational Intervention for COVID-19 Misinformation Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Jon Agley, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Indiana_CTSI_Agley_2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: COVID19 Behavioral Prophylaxis
Keywords: misinformation; trust; prevention
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Although this is, in practice, a double-blind study since participants will be unaware that they are randomized and all study mechanics will be processed by computer, analysts will not be blinded to the meaning of the assignment variable. However, two independent consultant analysts have been retained to verify all results and subsequent interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention arm (Experimental): The primary intervention in this study will be an infographic that is designed to build trust in the scientific process (as described in the Intervention section). This arm will introduce the intervention and then instruct the participant to review it carefully (including a mandated pause on the infographic screen) before continuing to the remaining data collection.
  Interventions: Behavioral: Brief informational infographic
- Placebo Control arm (Placebo Comparator): The comparator in this study will be a control ("placebo") infographic that is completely unrelated to science (As described in the Placebo Control section). This arm will introduce the control infographic and then instruct the participant to review it carefully (including a mandated pause on the infographic screen) before continuing to the remaining data collection.
  Interventions: Behavioral: Placebo control (non-behavioral infographic)

INTERVENTIONS:
Behavioral: Brief informational infographic — The primary intervention in this study will be an infographic that is designed to build trust in the scientific process. Infographics are preferable to narratives or text because they center visuals as part of the storytelling process and facilitate cognitive information processing, knowledge absorption, and enhanced persuasion. The study's infographic design will follow best practices in health communication. The message will be simple and jargon free. Visuals will include individuals (scientists), charts, text, and numbers. Attention will be paid to images, color, frames, representation, and composition (e.g., how the elements in the infographic are organized to show their relationship to each other).
  Arms: Brief Intervention arm
Behavioral: Placebo control (non-behavioral infographic) — The comparator in this study will be a control ("placebo") infographic that is completely unrelated to science (e.g., about cats), but that is developed using the same communication and graphical style.
  Arms: Placebo Control arm

SUMMARY:
As the coronavirus disease 2019 (COVID-19) pandemic has continued to affect life in the United States, the important role of non-pharmaceutical preventive behaviors (such as wearing a face mask) in reducing harm has become clear. In parallel to the pandemic, researchers have observed an "infodemic" of misinformed or inconsistent narratives about COVID-19. There is growing evidence that misinformed COVID-19 narratives are associated with a wide variety of undesirable behavior (e.g., burning down cell towers). Further, individuals' adherence to recommended COVID-19 preventive guidelines has been inconsistent, and such mandates have engendered opposition and controversy. Recent research suggests the possibility that trust in science and scientists may be an important thread to weave throughout these seemingly disparate components of the modern public health landscape. Thus, this paper describes the protocol for a randomized trial of a brief, digital intervention to increase trust in science.

The objective of this trial is to examine if exposure to a curated infographic can increase trust in science, reduce believability of misinformed narratives, and increase likelihood to engage in preventive behaviors.

DETAILED DESCRIPTION:
The investigators propose a single-stage, randomized, superiority trial with 2 parallel groups allocated with a 1:1 ratio. The comparator in this study will be a control ("placebo") infographic that is completely unrelated to science (e.g., about cats), but that is developed using the same communication and graphical style.

Subjects will be recruited using the Prolific data collection platform, which is one of two primary online crowdsourced research platforms (the other is Amazon's Mechanical Turk, or mTurk).

To be included, participants must be identified by Prolific as part of a nationally-representative sample. Participants will also be required to be age 18 or older, and to reside in the United States. Individuals who decline to digitally sign the informed consent document will be excluded and replaced. Per recent best practice recommendations for crowdsourced digital research, attention checks and screens for "bots" and international users with virtual private networks to mimic US IP addresses will be embedded within the instruments, and failure of more than one attention check, or any bot/location check will result in subject exclusion and replacement. Replacements will be drawn in such a way as to preserve the representativeness of the sample.

Missing data will be addressed using either full information maximum likelihood or Markov Chain Monte Carlo multiple imputation strategies. When there is a violation of missing at random (which is unlikely) in preliminary analyses, the investigators will incorporate strategies representing the missingness. The researchers will further explore data quality in terms of outliers, measurement error, non-normality, and variance heterogeneity. Robust methods of analysis (e.g., Huber-White robust standard errors) will be used, as appropriate. For all multi-item measures, reliability will be evaluated prior to computation of the variable.

ELIGIBILITY:
Inclusion Criteria:

* To be included, participants must be identified by Prolific as part of a nationally-representative sample. Participants will also be required to be age 18 or older, and to reside in the United States.

Exclusion Criteria:

* Individuals who decline to digitally sign the informed consent document will be excluded and replaced. Per recent best practice recommendations for crowdsourced digital research, attention checks and screens for "bots" and international users with virtual private networks to mimic US internet protocol addresses will be embedded within the instruments, and failure of more than one attention check, or any bot/location check will result in subject exclusion and replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1017 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in trust in science | Pre-intervention and immediately post-intervention
  21-item scale developed by Nadelson et al [1] called the Trust in Science Inventory. It is scored from 1 to 5, where 1 indicates low trust and 5 indicates high trust.
Believability profiles | Immediately post-intervention
  Will be computed using latent profile analysis of believability measures. These measures were developed and first used in our recent study of COVID-19 narratives [2]. Response options for these measures used well-established semantic differential responses for believability of different statements (e.g., as in Herzberg et al.) [3] ranging from [1: Extremely unbelievable] to [7: Extremely believable]. Exact measures used to generate profiles for this study will be available in the published protocol paper (to be submitted).
Preventive behavioral intentions | Immediately post-intervention
  A series of six questions based on the US Centers for Disease Control and Prevention's recommended COVID-19 preventive behaviors. [4] Questions will be written according to Azjen's guide to intention questionnaires [5].

OTHER OUTCOMES:
Political orientation (covariate 1) | Immediately post-intervention
  Scale variable (0: Conservative to 10: Liberal) as in our prior work [2, 6]
Religious commitment (covariate 2) | Immediately post-intervention
  Scale variable (0: Low commitment to 10: High commitment) as in our prior work [2, 6]
Sociodemographics (covariates 3 through 6) | Immediately post-intervention
  Race/ethnicity, gender, age, and education level using standardized questions
COVID-19 diagnosis (covariates 7 and 8) | Immediately post-intervention
  Two self report questions. The first asks whether the respondent has been diagnosed with COVID-19, and the second asks more broadly whether the respondent believes they have had COVID-19. Question wording will be per Bruine de Bruin (2020) [7].
Perceived severity of COVID-19 (covariate 9) | Immediately post-intervention
  Based on the Health Belief Model as used in Yıldırıma & Gülerc [8].
Self-efficacy to act regarding COVID-19 | Immediately post-intervention
  Based on the Health Belief Model as used in Yıldırıma & Gülerc [8].
Normative beliefs about friends' and family's COVID-19 behaviors | Immediately post-intervention
  Single item from Chambon et al [9].

CONTACTS AND LOCATIONS:
Locations (1):
- Digital Intervention (Prolific Study Panel), Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified data (full dataset) will be made available along with the publication of the primary results paper from this study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Fully de-identified data will be made available along with the publication of the primary results paper from this study.

REFERENCES:
- [Background] Nadelson L, Jorcyk C, Yang D, et al. I just don't trust them: The development and validation of an assessment instrument to measure trust in science and scientists. School Science and Mathematics. 2014;114(2):76-86.
- [Background] Agley J, Xiao Y. Existence of differential belief profiles of COVID-19 narratives: The role of trust in science. Research Square. 2020;Preprint.
- [Background] Herzberg KN, Sheppard SC, Forsyth JP, Crede M, Earleywine M, Eifert GH. The Believability of Anxious Feelings and Thoughts Questionnaire (BAFT): a psychometric evaluation of cognitive fusion in a nonclinical and highly anxious community sample. Psychol Assess. 2012 Dec;24(4):877-91. doi: 10.1037/a0027782. Epub 2012 Apr 9. PMID 22486595
- [Background] CDC. How to protect yourself & others. Centers for Disease Control and Prevention. https://www.cdc.gov/coronavirus/2019-ncov/prevent-getting-sick/prevention.html. Published 2020. Accessed July 17, 2020.
- [Background] Ajzen I. Theory of planned behavior questionnaire. Measurement Instrument Database for Social Science. https://www.midss.org/sites/default/files/tpb.construction.pdf. Published 2013. Accessed July 17, 2020.
- [Background] Agley J. Assessing changes in US public trust in science amid the COVID-19 pandemic. Public Health. 2020 Jun;183:122-125. doi: 10.1016/j.puhe.2020.05.004. Epub 2020 May 13. PMID 32405095
- [Background] Bruine de Bruin W. Age Differences in COVID-19 Risk Perceptions and Mental Health: Evidence From a National U.S. Survey Conducted in March 2020. J Gerontol B Psychol Sci Soc Sci. 2021 Jan 18;76(2):e24-e29. doi: 10.1093/geronb/gbaa074. PMID 32470120
- [Background] Yildirim M, Guler A. COVID-19 severity, self-efficacy, knowledge, preventive behaviors, and mental health in Turkey. Death Stud. 2022;46(4):979-986. doi: 10.1080/07481187.2020.1793434. Epub 2020 Jul 16. PMID 32673183
- [Background] Chambon M, Dalege J, Elberse JE, Harreveld Fv. A psychological network approach to factors related to preventive behaviors during pandemics: A European COVID-19 study. PsyArXiv. 2020:https://doi.org/10.31234/osf.io/es31245v.
- [Derived] Agley J, Xiao Y, Thompson EE, Chen X, Golzarri-Arroyo L. Intervening on Trust in Science to Reduce Belief in COVID-19 Misinformation and Increase COVID-19 Preventive Behavioral Intentions: Randomized Controlled Trial. J Med Internet Res. 2021 Oct 14;23(10):e32425. doi: 10.2196/32425. PMID 34581678
- [Derived] Agley J, Xiao Y, Thompson EE, Golzarri-Arroyo L. COVID-19 Misinformation Prophylaxis: Protocol for a Randomized Trial of a Brief Informational Intervention. JMIR Res Protoc. 2020 Dec 7;9(12):e24383. doi: 10.2196/24383. PMID 33175694